CLINICAL TRIAL: NCT03659526
Title: Development, Validation and Implementation of a New Quantitative Stress Echocardiographic Test for Myocardial Ischaemia
Brief Title: Quantitative Stress Echocardiography to Diagnose Myocardial Ischaemia
Acronym: DEVISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Wales (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Universitat Pompeu Fabra (Other); Hull University Teaching Hospitals NHS Trust (Other Government); Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Professor Alan G Fraser, Professor of Cardiology, University Hospital of Wales
Other Study IDs: IRAS Project ID 136434
Record Dates: First submitted 2018-08-17; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Ischemia, Myocardial
Keywords: Myocardial velocity imaging; Strain; Strain rate; Speckle tracking; Deformation; Quantitative; Echocardiography; Machine learning
MeSH Terms: conditions — Myocardial Ischemia; Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Healthy volunteers or if they have had normal invasive or CT coronary arteriography or other functional imaging test
  Interventions: Diagnostic Test: Deformation imaging
- Deformation imaging: Significant coronary disease (diameter stenosis >50%) has been diagnosed on arteriography or on CT angiography. Fractional flow reserve will be measured as the reference criterion.
  Interventions: Diagnostic Test: Deformation imaging
- High p(CAD): Intermediate-to-high probability of significant epicardial coronary disease (>50%).
  Interventions: Diagnostic Test: Deformation imaging
- All comers: Probability of severe disease ranging from 15 to 85%.
  Interventions: Diagnostic Test: Deformation imaging

INTERVENTIONS:
Diagnostic Test: Deformation imaging — Deformation parameters derived using myocardial velocity imaging or speckle tracking

SUMMARY:
Patients with chest pain on exertion need a reliable non-invasive test to identify if they have inducible myocardial ischaemia. This would reduce the use of diagnostic coronary arteriography, avoid its risks and costs, and guide clinical decisions. Conventional stress echocardiography has poor reproducibility because it relies on qualitative and subjective interpretation. Quantitative approaches based on precise and reliable measurements of myocardial velocity, strain, strain rate and global longitudinal strain have been shown to be able to accurately diagnose myocardial ischaemia. A more accurate test using myocardial velocity imaging was not implemented by ultrasound vendors although it provided an objective measurement of myocardial functional reserve on a continuous scale from normality to severe ischaemia.

The investigators propose an original approach to create a diagnostic software tool that can be used in routine clinical practice. The investigators will extract and compare quantitative data obtained through myocardial velocity imaging and speckle tracking in subjects who undergo dobutamine stress echocardiography.

The data will be analysed using advanced computational mathematics including multiple kernel learning and joint statistics applied to multivariate data across multiple dimensions (including velocity, strain and strain rate traces). This approach will be validated against quantitative coronary arteriography and fractional flow reserve. The results will be displayed as parametric images and placed into a reporting tool. The output will determine the presence and severity of myocardial ischaemia. These new tools will have the capacity for iterative learning so that the precision of the diagnostic conclusions can be continuously refined.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain, chest pain equivalent

Exclusion Criteria:

* acute coronary syndrome with elevated troponin, severe heart valve disease, uncontrolled hypertension (resting SBP >200mmHg), cardiomyopathy, contraindication to dobutamine, pregnancy

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Secondary care referrals
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2016-01-21 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of quantitative measures of dobutamine stress echocardiography | 18 months
  Echocardiographic measurements of segmental myocardial velocity, strain, strain rate and wall motion scoring referenced against measurements derived from coronary angiography.

SECONDARY OUTCOMES:
Lowest dose of dobutamine to provoke measurable marker of inducible myocardial ischaemia | 18 months
  Using modelling techniques applied predict lowest dose of dobutamine to maintain diagnostic accuracy
Diagnostic accuracy of using machine learning to interpret multiparametric and multidimensional datasets to diagnose myocardial ischaemia | 18 months
  Use modelling to combine pre-test probabilities (based on risk factors such as age), physiological factors (e.g., heart rate) that are associated with longitudinal function and data derived throughout the cardiac cycle (i.e., based on analysis of velocity or strain curves and not just a single value like peak velocity or strain).

CONTACTS AND LOCATIONS:
Overall Officials: Alan G Fraser, Principal Investigator — University Hospital Wales
Locations (4):
- UZ Leuven, Leuven, Belgium
- Danderyd Hospital, Stockholm, Sweden
- United Kingdom (2):
  - University Hospital Wales, Cardiff
  - Castle Hill Hospital, Cottingham

IPD SHARING:
Plan to Share IPD: Undecided